CLINICAL TRIAL: NCT04671225
Title: Psychoeducation for Patients With Bipolar Disorder in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Rwanda (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUUR2020DKRW
Record Dates: First submitted 2020-11-24; First posted 2020-12-17 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2020-11

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: The RCT: Outpatients from the two-referral hospitals in Rwanda will be invited to participate and be allocated to the intervention group or waiting list.
  The district trial: This trial compares the impact of the intervention given at the district level with the intervention conducted at the referral hospital.
  Randomization:
  Study participants at the hospital level who meet the inclusion criteria and sign the informed consent form will be randomized individually into either intervention-arm or waiting list through block-randomization with a ratio of 1:1.
  Patients at the district level will not be randomized since we are unsure of the number of patients with Bipolar Disorder at these levels fearing that the sample size will be too small. Instead, all will be offered participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Psychoeducation at the referral hospital (Experimental): Intervention: Manual-structured group psychoeducation.
  Interventions: Behavioral: Groups Psychoeducation
- Waiting list - at the referral hospital (Other): Participants in the control group will be assigned to a waiting list and receive group-psychoeducation after the active intervention groups.
  Interventions: Behavioral: Waiting-list

INTERVENTIONS:
Behavioral: Groups Psychoeducation — Manual-structured group psychoeducation with 8 sessions of 90 minutes over the course of 8 weeks (at one session per week). The manual is centred on behavioural principles from social education and self-regulation philosophies. All groups will have 6-8 participants and two health professionals to conduct the sessions; a psychiatric nurse and either a psychologist or a psychiatric resident. Patients will be offered to invite their relatives for 2-3 psychoeducation-days for relatives.
  Arms: Intervention - Psychoeducation at the referral hospital
Behavioral: Waiting-list — Participants in the control group will be assigned to a waiting list and receive group-psychoeducation after the active intervention groups.
  Arms: Waiting list - at the referral hospital

SUMMARY:
Background: Mental health- and neurological disorders constitute 13% of the global burden of disease. Alarmingly this burden has risen by 41% in the last 20 years. In low-and-middle-income countries as few as 10% of people living with bipolar disorder receive care. In western countries, the efficacy of psychoeducation, as an add-on treatment to pharmacotherapy in the treatment of symptoms and in relapse prevention initiatives with respect to bipolar disorder, is well documented. Yet, few studies on psychosocial interventions for bipolar disorder have been conducted in a low-income country.

Aim: To determine the effect, feasibility and acceptability of psychoeducation for patients with bipolar disorder on all three levels of the health care system in Rwanda - at the community health centre, district- and university hospital.

Methods: Patients will be randomized into either group A) group-psychoeducation at a referral hospital; or B) group-psychoeducation for both patients and relatives or C) waiting list. Moreover a district trial will test the impact and feasibility of psychoeducation at the district level.

Outcomes: Reduction in symptom severity and incidence of relapse, improved quality of life, medical adherence and knowledge, as well as reduced self-stigmatization.

Perspectives: If proven successful, this is of importance for closing the huge treatment gap in mental health particularly affecting low- and middle-income countries and may reduce the mortality and increase quality of life in the population suffering from bipolar disorder. Furthermore, potential positive outcomes may be implemented in similar low-resource settings elsewhere.

DETAILED DESCRIPTION:
Background: Mental health and neurological disorders constitute 13% of the global burden of diseases. Alarmingly this burden has risen by 41% in the last 20 years. It is estimated that severe mental disorders (i.e. severe depression, bipolar disorder, schizophrenia and other psychotic disorders) have a two to three times higher average mortality compared to the general population. Treatment rates for these disorders are low in low-and-middle-income countries (LMICs), where treatment gaps of more than 90% have been documented.

In western countries, the efficacy of psychoeducation, as an add-on treatment to pharmacotherapy in the treatment of symptoms and relapse prevention initiatives concerning bipolar disorder (BD), is well documented. Yet, few studies on psychosocial interventions for BD have been conducted in low-income countries.

The overall aim of the study is to determine the effect, feasibility and acceptability of psychoeducation for patients with BD in Rwanda.

Methods: The study is divided into a prospective randomized controlled trial (RCT) and a district trial. Patients with bipolar disease type I or II that meet DSM-V diagnostic criteria given by a trained psychiatrist and age ≥ 18 years will be invited to participate.

For the RCT study participants will be randomised to 1) group-psychoeducation for patients and relatives, 2) a waiting list. The RCT will take place at a referral hospital. The district trial compares the impact of psychoeducation given at the district level by mental health nurses with psychoeducation conducted at referral hospitals.

Intervention: Manual-structured group psychoeducation with eight sessions of 90 minutes over eight weeks (at one session per week). Patients will be offered to invite their relatives for 2-3 psychoeducation-days for relatives.

Outcomes: The primary outcome is a reduction in symptom severity, the incidence of relapse and hospitalization. Secondary outcomes include Improved quality of life and medication adherence and knowledge, as well as reduced self-stigmatization. All outcomes will be assessed at baseline, immediately post-intervention, and at the 3 and 6 months follow-up.

Sample size: In the literature on group-psychoeducation, 13 out of 18 RCT's have a reduction in general psychiatric symptom severity, the incidence of relapse and hospitalization as main outcomes. Eighteen RCT's on group psychoeducation for BD were reviewed before a study of Colom et al. was selected as the base of the power calculation. The incidence of relapse in the study was (92%) (55 subjects) in the control group vs 67% (40 subjects) in the psychoeducation group. For this study, a sample size of 40 patients for each arm is required to achieve a level of 80% power with a 5% level of significance when comparing the mean change in each intervention with the control arm via a two-sample t-test. Adjusting for a drop-out rate of 20%: 40/(1-(20/100))= 50 participants will be needed for each group (50 for intervention, 50 for waiting-list and 50 for the district trial).

Randomization: Study participants at the hospital level who meet the inclusion criteria and sign the informed consent form will be randomized individually into either intervention-arm or waiting list through block-randomization with a ratio of 1:1.

Patients at the district level will not be randomized since the number of patients with BD at these levels is unknown and can result in the sample size will be too small. Instead, all will be offered participation.

Ethical Approval The research protocol and study-related documents have been approved by the College of Medicine and Health Sciences Institutional Review Board, Rwanda and The National Council for Science and Technology (NCST) in Rwanda.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of BD type I or II that meets DSM-V diagnostic criteria given by a trained psychiatrist
* No episode in the preceding 4 weeks. Age ≥ 18 years.

Exclusion Criteria:

* Previous participation in any structured psychological intervention
* Insufficient understanding of Kinyarwanda
* Clinical evidence of substantial cognitive impairments.
* Alcohol or drug-dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients that relapse | 1 year
  Relapse is defined as a new mood episode of mania (scores above or equal to 20 on the Young Mania Rating Scale (YMRS)(25)), hypomania (above or equal to 12 on the YMRS), or depression (above or equal to 17 on the Hamilton Depression Scale- 17(HDRS-17(26)) or mixed episode (above or equal to 20 on the YMRS and 12 on the HDRS- 17).

SECONDARY OUTCOMES:
Number of patient reporting improvement in medical adherence | 1 year
  Medication Adherence Rating Scale (MARS) will be used to assess beliefs and barriers to medication adherence. Total scores on the MARS may range between 0 and 10, with a higher score indicating better medication adherence.
Number of patient reporting reduction in self-stigma | 1 year
  Internalized Stigma of Mental Illness Inventory - 9-item Version (ISMI-9) will be used to assess self-stigma. The resulting score should range from 1 to 4. A score ranging between 1.00-2.50: does not report high internalized stigma vs. a score ranging between 2.51-4.00: indicating high internalized stigma
Improvement of illness severity | 1 year
  The Clinical Global Impression (CGI-I /CGI-S) will be used for the clinicians to assess how much the participant's condition has improved. The first scale: CGI-Severity (CGI-S) rates illness severity at baseline. The score range between 1 and 7with a higher score indicating serve illness.
  The other scale CGI-Improvement (CGI-I) tracks improvement after initiation of treatment on a scale from 1 to 7. Four indicates no change. A low score indicates improvement and a high score of worsening symptoms.
Acceptability of the intervention | 1 year
  A seven-item questionnaire based on The theoretical framework of acceptability will be used to access the acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Per Kallestrup, Prof., Study Chair — University of Aarhus
Locations (2):
- Rwanda (2):
  - Ndera Hospital, Kigali
  - The University Teaching Hospital of Kigali (CHUK), Kigali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vigo D, Thornicroft G, Atun R. Estimating the true global burden of mental illness. Lancet Psychiatry. 2016 Feb;3(2):171-8. doi: 10.1016/S2215-0366(15)00505-2. PMID 26851330
- [Background] Whiteford HA, Ferrari AJ, Degenhardt L, Feigin V, Vos T. The global burden of mental, neurological and substance use disorders: an analysis from the Global Burden of Disease Study 2010. PLoS One. 2015 Feb 6;10(2):e0116820. doi: 10.1371/journal.pone.0116820. eCollection 2015. PMID 25658103
- [Background] Gilbert BJ, Patel V, Farmer PE, Lu C. Assessing development assistance for mental health in developing countries: 2007-2013. PLoS Med. 2015 Jun 2;12(6):e1001834. doi: 10.1371/journal.pmed.1001834. eCollection 2015 Jun. PMID 26035429
- [Background] Rathod S, Pinninti N, Irfan M, Gorczynski P, Rathod P, Gega L, Naeem F. Mental Health Service Provision in Low- and Middle-Income Countries. Health Serv Insights. 2017 Mar 28;10:1178632917694350. doi: 10.1177/1178632917694350. eCollection 2017. PMID 28469456
- [Background] Mackenzie J, Kesner C. Mental health funding and the SDGs What now and who pays ? 2016;(May).
- [Background] Kleinman A. Global mental health: a failure of humanity. Lancet. 2009 Aug 22;374(9690):603-4. doi: 10.1016/s0140-6736(09)61510-5. No abstract available. PMID 19708102
- [Background] Liu NH, Daumit GL, Dua T, Aquila R, Charlson F, Cuijpers P, Druss B, Dudek K, Freeman M, Fujii C, Gaebel W, Hegerl U, Levav I, Munk Laursen T, Ma H, Maj M, Elena Medina-Mora M, Nordentoft M, Prabhakaran D, Pratt K, Prince M, Rangaswamy T, Shiers D, Susser E, Thornicroft G, Wahlbeck K, Fekadu Wassie A, Whiteford H, Saxena S. Excess mortality in persons with severe mental disorders: a multilevel intervention framework and priorities for clinical practice, policy and research agendas. World Psychiatry. 2017 Feb;16(1):30-40. doi: 10.1002/wps.20384. PMID 28127922
- [Background] Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ. 2004 Nov;82(11):858-66. Epub 2004 Dec 14. PMID 15640922
- [Background] Sankoh O, Sevalie S, Weston M. Mental health in Africa. Lancet Glob Health. 2018 Sep;6(9):e954-e955. doi: 10.1016/S2214-109X(18)30303-6. No abstract available. PMID 30103990
- [Background] Burns JK, Tomita A. Traditional and religious healers in the pathway to care for people with mental disorders in Africa: a systematic review and meta-analysis. Soc Psychiatry Psychiatr Epidemiol. 2015 Jun;50(6):867-77. doi: 10.1007/s00127-014-0989-7. Epub 2014 Dec 12. PMID 25515608
- [Background] Keynejad RC, Dua T, Barbui C, Thornicroft G. WHO Mental Health Gap Action Programme (mhGAP) Intervention Guide: a systematic review of evidence from low and middle-income countries. Evid Based Ment Health. 2018 Feb;21(1):30-34. doi: 10.1136/eb-2017-102750. Epub 2017 Sep 13. PMID 28903977
- [Background] Patel V. Global mental health: from science to action. Harv Rev Psychiatry. 2012 Jan-Feb;20(1):6-12. doi: 10.3109/10673229.2012.649108. PMID 22335178
- [Background] Colom F. The evolution of psychoeducation for bipolar disorder: from lithium clinics to integrative psychoeducation. World Psychiatry. 2014 Feb;13(1):90-2. doi: 10.1002/wps.20091. No abstract available. PMID 24497258
- [Background] Soo SA, Zhang ZW, Khong SJ, Low JEW, Thambyrajah VS, Alhabsyi SHBT, Chew QH, Sum MY, Sengupta S, Vieta E, McIntyre RS, Sim K. Randomized Controlled Trials of Psychoeducation Modalities in the Management of Bipolar Disorder: A Systematic Review. J Clin Psychiatry. 2018 May/Jun;79(3):17r11750. doi: 10.4088/JCP.17r11750. PMID 29727072
- [Background] Demissie M, Hanlon C, Birhane R, Ng L, Medhin G, Fekadu A. Psychological interventions for bipolar disorder in low- and middle-income countries: systematic review. BJPsych Open. 2018 Aug 30;4(5):375-384. doi: 10.1192/bjo.2018.46. eCollection 2018 Sep. PMID 30202599
- [Background] Aubry JM, Charmillot A, Aillon N, Bourgeois P, Mertel S, Nerfin F, Romailler G, Stauffer MJ, Gex-Fabry M, de Andres RD. Long-term impact of the life goals group therapy program for bipolar patients. J Affect Disord. 2012 Feb;136(3):889-94. doi: 10.1016/j.jad.2011.09.013. Epub 2011 Oct 5. PMID 21975136
- [Background] Simon GE, Ludman EJ, Unutzer J, Bauer MS, Operskalski B, Rutter C. Randomized trial of a population-based care program for people with bipolar disorder. Psychol Med. 2005 Jan;35(1):13-24. doi: 10.1017/s0033291704002624. PMID 15842025
- [Background] Bauer MS, McBride L, Williford WO, Glick H, Kinosian B, Altshuler L, Beresford T, Kilbourne AM, Sajatovic M; Cooperative Studies Program 430 Study Team. Collaborative care for bipolar disorder: part I. Intervention and implementation in a randomized effectiveness trial. Psychiatr Serv. 2006 Jul;57(7):927-36. doi: 10.1176/ps.2006.57.7.927. PMID 16816276
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Eaton J, McCay L, Semrau M, Chatterjee S, Baingana F, Araya R, Ntulo C, Thornicroft G, Saxena S. Scale up of services for mental health in low-income and middle-income countries. Lancet. 2011 Oct 29;378(9802):1592-603. doi: 10.1016/S0140-6736(11)60891-X. Epub 2011 Oct 16. PMID 22008429
- [Background] Colom F, Vieta E, Martinez-Aran A, Reinares M, Goikolea JM, Benabarre A, Torrent C, Comes M, Corbella B, Parramon G, Corominas J. A randomized trial on the efficacy of group psychoeducation in the prophylaxis of recurrences in bipolar patients whose disease is in remission. Arch Gen Psychiatry. 2003 Apr;60(4):402-7. doi: 10.1001/archpsyc.60.4.402. PMID 12695318
- [Background] Schriver M, Cubaka VK, Kyamanywa P, Cotton P, Kallestrup P. Twinning Ph.D. students from south and north: towards equity in collaborative research. Educ Prim Care. 2015 Sep;26(5):349-52. doi: 10.1080/14739879.2015.1079970. Epub 2015 Sep 21. No abstract available. PMID 26808804
- [Derived] Arnbjerg CJ, Musoni-Rwililiza E, Rurangwa NU, Bendtsen MG, Murekatete C, Gishoma D, Carlsson J, Kallestrup P. Effectiveness of structured group psychoeducation for people with bipolar disorder in Rwanda: A randomized open-label superiority trial. J Affect Disord. 2024 Jul 1;356:405-413. doi: 10.1016/j.jad.2024.04.071. Epub 2024 Apr 18. PMID 38640974
- [Derived] Arnbjerg CJ, Musoni-Rwililiza E, Rurangwa NU, Bendtsen MG, Murekatete C, Gishoma D, Carlsson J, Kallestrup P. Help-seeking patterns and level of care for individuals with bipolar disorder in Rwanda. PLOS Glob Public Health. 2023 Oct 10;3(10):e0002459. doi: 10.1371/journal.pgph.0002459. eCollection 2023. PMID 37815957
- [Derived] Musoni-Rwililiza E, Arnbjerg CJ, Murekatete C, Carlsson J, Kallestrup P, Gishoma D. Group psychoeducation for persons with bipolar disorder in Rwanda: a study protocol for a randomized controlled trial. Trials. 2022 Dec 2;23(1):971. doi: 10.1186/s13063-022-06926-1. PMID 36461128
- See also: WHO. Global Health Estimates 2016: Burden of disease by cause, age, sex, by country and by region, 2000-2016. 2018. — https://www.who.int/data/gho/data/themes/mortality-and-global-health-estimates

DOCUMENTS (1):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT04671225/Prot_000.pdf